CLINICAL TRIAL: NCT05149872
Title: Recovery of Carotid Body Function After Full Recovery Neuromuscular Block
Brief Title: The Breath-2 Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Martijn Boon, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: P21.083
Record Dates: First submitted 2021-11-09; First posted 2021-12-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Chemosensitivity
MeSH Terms: interventions — Muscle Relaxation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- spontaneous recovery (Other): Spontaneous recovery
  Interventions: Other: Muscle relaxation
- reversal with sugammadex 2 mg/kg (Other): reversal with sugammadex 2 mg/kg
  Interventions: Other: Muscle relaxation; Other: Reversal
- reversal with sugammadex 4 mg/kg (Other): reversal with sugammadex 4 mg/kg
  Interventions: Other: Muscle relaxation; Other: Reversal

INTERVENTIONS:
Other: Muscle relaxation — Rocuronium will be used to induce partial paralysis
Other: Reversal — Sugamamdex will be used to reverse muscle relaxation
  Arms: reversal with sugammadex 2 mg/kg; reversal with sugammadex 4 mg/kg

SUMMARY:
This is a randomized, cross over, experimental trial in which carotid body function will be evaluated in 35 healthy subjects during partial muscle relaxation and after recovery from muscle relaxation

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years

Exclusion Criteria:

* BMI index > 30 kg/m2
* Known or suspected neuromuscular disorders impairing neuromuscular function;
* Allergies to muscle relaxants, anesthetics or narcotics;
* A (family) history of malignant hyperthermia or any other muscle disease;
* Any neurological or psychiatric illness (including a history of anxiety).
* ASA class 3 or higher
* Gastro-oesophageal regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Carotid body function after full recovery of neuromuscular block | 40 minutes after full recovery of neuromuscular block
  Carotid body function will be determined by measuring acute hypoxic ventilatory response

SECONDARY OUTCOMES:
Carotid body function at symptomatic neuromuscular block | 5 minutes after stable partial neuromuscular block
  Carotid body function will be determined by measuring acute hypoxic ventilatory response
Carotid body function at full recovery of NMB symptoms | 0 minutes after full recovery of neuromuscular block symptoms
  Carotid body function will be determined by measuring acute hypoxic ventilatory response
Carotid body function after full recovery of neuromuscular block | 20 minutes after full recovery of neuromuscular block symptoms
  Carotid body function will be determined by measuring acute hypoxic ventilatory response
Carotid body function after full recovery of neuromuscular block | 40 minutes after full recovery of neuromuscular block symptoms
  Carotid body function will be determined by measuring acute hypoxic ventilatory response

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden Medical University, Leiden, South Holland, Netherlands